CLINICAL TRIAL: NCT06344819
Title: Acupuncture to Improve Outcomes in Sepsis Patient: The ACTIONS Trial
Brief Title: An Acupuncture Study for People At High Risk for Sepsis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-062
Record Dates: First submitted 2024-03-21; First posted 2024-04-03 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Sepsis
Keywords: sepsis; acupuncture; Memorial Sloan Kettering Cancer Center; 24-062
MeSH Terms: conditions — Sepsis | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Procedure: Acupuncture
- Sham Acupuncture (Sham Comparator)
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture involves insertion of thin filiform needles (gauze 30-40) at certain points on the body.
  Arms: Acupuncture
Other: Sham Acupuncture — During sham acupuncture, the point on the participant's thigh 6 inches proximal to the ST36 acupuncture point is gently tapped with an acupuncture needle guide tube and an acupuncture needle is taped flat to the skin. This point is not on any acupuncture meridian or point.
  Arms: Sham Acupuncture

SUMMARY:
Researchers think acupuncture may improve outcomes for participants with sepsis, based on laboratory studies and previous studies in people with sepsis. The purpose of this study to see whether real acupuncture can improve outcomes for participants with sepsis when compared to sham acupuncture. Sham acupuncture is performed the same way as real acupuncture but will use different needles and target different sites or places on the body than real acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Having MSK sepsis order-set placed within the previous 48 hours

Exclusion Criteria:

* The study Principal Investigator will review the medical record again prior to enrollment to exclude non-sepsis patients (Even though the placement of sepsis order set already screens out such patients, subsequent clinical development after sepsis order set placement may generate new information that deems the patient not septic.)
* Admitted to ICU before being approached for consenting
* Having an implanted medical device, such as a pacemaker or implantable cardioverter-defibrillator (ICD), with which electroacupuncture
* Unable to obtain informed consent due to a participant's mental status and absence of an individual authorized to give consent on the participant's behalf
* The patient is on an interventional clinical trial and its Principal Investigator does not give approval to enrollment to this study (e.g. genomic profiling, biospecimen, or observational studies do not require PI approval).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-03-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited compared to the number of participants who complete study treatment. | Up to 2 years
  To assess the feasibility of conducting a randomized controlled trial of acupuncture in hospitalized patients who are at risk for sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Deng, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org